CLINICAL TRIAL: NCT05897788
Title: Text-Messaging Telehealth and Contingency Management for Opioid Use Disorder Treatment Engagement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, M. Kit Delgado, MD, Assistant Professor of Emergency Medicine and Epidemiology, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 853153
Record Dates: First submitted 2023-05-23; First posted 2023-06-09 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder; Opioid Dependence With Current Use (Disorder)
Keywords: Opioid use disorder; Contingency Management; text-based interventions
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Patients enrolled into the Way to Health CareConnect text line as part of usual care and meeting eligibility criteria will be enrolled in this randomized control trial and randomized to: Augmented usual care, standard Way to Health CareConnect text line Patients can call or text the on-call substance use navigators (SUN) from 9a-9p, 7 days a week. Augmented usual care + text-message check-ins, standard Way to Health CareConnect Text line Patients can call or text the on-call substance use navigators (SUN) from 9a-9p, 7 days a week AND (text-message check-ins) patients will receive automated text-message check-ins up to once per day for 30 days to see if the patient needs help with anything.
  Augmented usual care + contingency management (standard Way to Health CareConnect Text line) and, participants will be compensated for going to their follow-up appointments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Augmented Usual Care (AUC) (No Intervention): AUC: Standard Way to Health Care text line. Patients can call or text the on-call substance use navigators (SUN) from 9a-9p, 7 days a week.
  Participants across all arms will receive an intake survey, and follow-up surveys at day 15, day 30, month 3, and month 6.
- Augmented usual care + text-message check-ins (Active Comparator): AUC: Standard Way to Health Care text line. Patients can call or text the on-call substance use navigators (SUN) from 9a-9p, 7 days a week.
  Text check-in: Patients will also receive incentives for engagement with treatment and
  Participants across all arms will receive an intake survey, and follow-up surveys at day 15, day 30, month 3, and month 6.
  Interventions: Behavioral: Text Message Check-ins
- Augmented Usual care + Contingency Management (CM) (Active Comparator): AUC: Standard Way to Health Care text line. Patients can call or text the on-call substance use navigators (SUN) from 9a-9p, 7 days a week.
  Participants across all arms will receive an intake survey, and follow-up surveys at day 15, day 30, month 3, and month 6.
  CM: Patients will also receive incentives for engagement with treatment.
  Interventions: Behavioral: Contingency Management
- Augmented usual care + text-message check-ins + contingency management (Active Comparator): AUC: Standard Way to Health Care text line. Patients can call or text the on-call substance use navigators (SUN) from 9a-9p, 7 days a week.
  Text check-in: Patients will also receive incentives for engagement with treatment and
  Participants across all arms will receive an intake survey, and follow-up surveys at day 15, day 30, month 3, and month 6.
  CM: Patients will also receive incentives for engagement with treatment.
  Interventions: Behavioral: Text Message Check-ins; Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Text Message Check-ins — Patients will receive automated text-message check-ins up to once per day for 30 days to see if the patient needs help with anything AND patients can call or text the on-call substance use navigators (SUN) from 9a-9p, 7 days a week.
  Arms: Augmented usual care + text-message check-ins; Augmented usual care + text-message check-ins + contingency management
Behavioral: Contingency Management — Patients will receive incentives for engagement with treatment. Participant will receive compensation for filling their buprenorphine scripts at discharge and attending their follow-up care appointments.
  Arms: Augmented Usual care + Contingency Management (CM); Augmented usual care + text-message check-ins + contingency management

SUMMARY:
There is growing recognition of the need for approaches to initiate treatment wherever patients touch the health care system, including the Emergency Department (ED). Most research has focused on initiation of medications for opioid use disorder (MOUDs) in the ED rather than ensuring continued treatment post-discharge. The investigators propose to adapt evidence-based interventions to support patients' complex needs and facilitate continued treatment, rather than discharging them and having them navigate outpatient treatment systems with limited support. The research team will randomize participants into 1 of 4 arms to receive varying degrees of augmented usual care, including daily check-ins and contingency management. The investigators plan to examine the effects of check-ins and contingency management on engagement with addiction treatment and equity of treatment effects among racial and ethnic subgroups and assess important moderators of treatment effects.

DETAILED DESCRIPTION:
The investigators are proposing to conduct a randomized controlled trial to determine the effectiveness of various text-based and contingency management interventions on Opioid Use Disorder patients. Our goals are to measure their engagement with recovery treatment. The research team plan to enroll 1,649 participants into one of the following 4 arms.

Patients enrolled into the Way to Health CareConnect text line as part of usual care and meeting eligibility criteria will be enrolled in this randomized control trial and randomized to:

Augmented usual care (standard Way to HealthCareConnect text line) Patients can call or text the on-call substance use navigators (SUN) from 9a-9p, 7 days a week.

Augmented usual care + text-message check-ins (standard Way to Health CareConnect Text line) Patients can call or text the on-call substance use navigators (SUN) from 9a-9p, 7 days a week AND (text-message check-ins) patients will receive automated text-message check-ins up to once per day for 30 days to see if the patient needs help with anything.

Augmented usual care + contingency management (standard Way to Health CareConnect Text line) and, participants will be compensated for going to their follow-up appointments.

Augmented usual care + CM + Text-message check-ins (standard Way to Health CareConnect text line) AND text-message check-ins-patients will receive automated text-message check-ins up to once per day for 30 days to see if the patient needs help with anything AND, participants will receive compensation for attending their follow-up appointments.

Patients enrolled in the trial will also be invited to complete the intake survey and follow-up surveys. Patients will receive financial compensation for completing these surveys. The study team plans to enroll 1,649 participants for this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 or older
* Screen positive for OUD
* Bridge buprenorphine prescription (emergency department (ED) enrollment - Buprenorphine prescription at ED discharge; Bridge clinic enrollment - new buprenorphine prescription associated with on-demand or drop-in encounter
* English reading ability
* Have a mobile phone capable of receiving text messages

Exclusion Criteria:

* Not being up to date with requirements above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1808 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Engagement in any addiction treatment at 30 days of randomization | 31 days
  Engagement in any addiction treatment within 30 days of randomization (measured on day 31)

SECONDARY OUTCOMES:
ED and Hospital Utilization and mortality | 6 months
  Subsequent ED and hospital utilization and mortality. The investigators have developed standardized data queries to capture all ED visits, hospitalizations, and mortality out to 6 months from enrollment. To capture encounters outside study health systems, the study team will obtain linked records from the regional health information exchanges (HIEs) - HealthShare Exchange for Penn and Cooper, Care Everywhere for Alameda). Will subsequently link the patient data to the National Death Index to capture of out-of-hospital mortality not captured in Electronic Health Records (EHRs) or HIEs.
Engagement in addition treatment within 14 days | 15 days
  Engagement in any addiction treatment within 14 days of randomization (measured on day 15)

OTHER OUTCOMES:
Comparative analysis across groups | 30 days
  For the exploratory outcomes at 30-days post-randomization, the investigators will use similar logistic regression models to compare the groups on enrollment and receipt of treatment, and on Urine Drug Screens (UDS) for illicit opioids. For ED visits and hospitalizations, the investigators will use zero-inflated negative binomial regression models if there is sufficient variability in these responses, and logistic regression models (for dichotomized versions of these responses) otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: Kit Delgado, MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT05897788/Prot_SAP_ICF_000.pdf